CLINICAL TRIAL: NCT01590602
Title: REGISTRY-JHD - an Observational Study of the European Huntington's Disease Network (EHDN)
Acronym: JHD
Status: Completed | Type: Observational
Sponsor: European Huntington's Disease Network (Network)
Responsible Party: Sponsor
Other Study IDs: REGISTRY-JHD
Record Dates: First submitted 2012-03-22; First posted 2012-05-03 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Huntington Disease, Juvenile
Keywords: Huntington's Disease; European Huntington's Disease Network; Juvenile HD; EHDN; REGISTRY
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- JHD cases: All ages included, but must have an HD age of onset 25 or below

SUMMARY:
The study aims to monitor the progression of symptoms and signs of those affected by JHD using modified UHDRS scales of motor and function (functional assessment, TFC). This will provide some basic data to analyse the usefulness of the proposed rating scales. Specifically, the initial aim is to assess these rating scales using an iterative process.

There may be significant delays in diagnosis of JHD especially if the young person presents with behavioural problems. Caregivers will be asked questions to capture the number of contacts with professionals in the time between onset of concerns about the young person and the confirmation of diagnosis.

Aim is to monitor the progression of symptoms and signs of those affected by JHD using modified UHDRS scales of motor and function (functional assessment, TFC). This will provide some basic data to analyse the usefulness of the proposed rating scales.

DETAILED DESCRIPTION:
Juvenile Huntington's disease (JHD), defined as motor symptom onset before 21 years of age, has been recognised as being at one end of the phenotypic spectrum of HD. In many studies the proportion of cases meeting this definition has varied, but it is usually less than 10% and more probably 5%.

At present, no treatment is available which will alter the natural history of the condition; however, there is considerable research activity being undertaken to identify novel treatments. Any new disease-modifying treatment will have to be evaluated in a clinical trial with a predetermined outcome measure. Given the relatively slow rate of progression of HD, such a trial may have to last several years and as a consequence be less attractive from a commercial perspective. Patients with JHD have more extensive pathology but are frequently excluded from clinical trials because of the differing phenotype; this study will assess the feasibility of using this rating scale; if it or a further modification can be used and is sensitive to disease progression over relatively short time periods, then it is likely to have a significant impact on study trial design and cost.

Given the rarity of JHD, wide collaboration of scientists, clinicians and families affected by JHD internationally is important. As might be expected, the pathology in JHD is more widespread. Therefore, we need the ability to assess treatments, which alter the natural history on this subgroup of patients.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of Juvenile-onset HD (motor onset as measured by TMS > 5, Diagnostic Confidence level = 4, AND age of onset aged 25 or younger).
* With family history of HD or DNA testing results demonstrating the presence of the HD mutation (i.e. a CAG repeat expansion within the HD gene >35 on larger allele).
* All participants must be able to provide consent for themselves, have a parent/guardian who can provide parental permission, or have an authorized legal representative who can provide consent.

Exclusion Criteria:

* Participants who are unable to understand the study protocol or unable to give informed consent, and have no legal representative.
* Age of onset ≥26

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HD patients of all ages with an age of onset below 26
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2011-11; Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Evalutation of assessments for HD | 5 years
  If the assessment used as in the study or further modified proofs to be sensitive to disease progression over relatively short time periods, then it is likely to have a significant impact on study trial design and cost.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Quarrell, MD, Principal Investigator — Sheffield Children's Hospital
Locations (2):
- University Hospital of Ulm, Dept. of Neurology, Ulm, Germany
- Sheffield Children's Hospital, Department of Clinical Genetics, Sheffield, United Kingdom

REFERENCES:
- [Background] Rickards H, De Souza J, van Walsem M, van Duijn E, Simpson SA, Squitieri F, Landwehrmeyer B; European Huntington's Disease Network. Factor analysis of behavioural symptoms in Huntington's disease. J Neurol Neurosurg Psychiatry. 2011 Apr;82(4):411-2. doi: 10.1136/jnnp.2009.181149. Epub 2010 Apr 14. PMID 20392980
- [Background] Orth M, Handley OJ, Schwenke C, Dunnett SB, Craufurd D, Ho AK, Wild E, Tabrizi SJ, Landwehrmeyer GB; Investigators of the European Huntington's Disease Network. Observing Huntington's Disease: the European Huntington's Disease Network's REGISTRY. PLoS Curr. 2010 Sep 28;2:RRN1184. doi: 10.1371/currents.RRN1184. PMID 20890398
- [Background] Orth M; European Huntington's Disease Network; Handley OJ, Schwenke C, Dunnett S, Wild EJ, Tabrizi SJ, Landwehrmeyer GB. Observing Huntington's disease: the European Huntington's Disease Network's REGISTRY. J Neurol Neurosurg Psychiatry. 2011 Dec;82(12):1409-12. doi: 10.1136/jnnp.2010.209668. Epub 2010 Nov 19. No abstract available. PMID 21097549
- [Background] Busse M, Al-Madfai DH, Kenkre J, Landwehrmeyer GB, Bentivoglio A, Rosser A; European Huntington's Disease Network. Utilisation of Healthcare and Associated Services in Huntington's disease: a data mining study. PLoS Curr. 2011 Jan 21;3:RRN1206. doi: 10.1371/currents.RRN1206. PMID 21304753
- [Background] Lopez-Sendon JL, Royuela A, Trigo P, Orth M, Lange H, Reilmann R, Keylock J, Rickards H, Piacentini S, Squitieri F, Landwehrmeyer B, Witjes-Ane MN, Jurgens CK, Roos RA, Abraira V, de Yebenes JG; European HD Network. What is the impact of education on Huntington's disease? Mov Disord. 2011 Jul;26(8):1489-95. doi: 10.1002/mds.23385. Epub 2011 Mar 22. PMID 21432905
- [Background] Ho AK, Hocaoglu MB; European Huntington's Disease Network Quality of Life Working Group. Impact of Huntington's across the entire disease spectrum: the phases and stages of disease from the patient perspective. Clin Genet. 2011 Sep;80(3):235-9. doi: 10.1111/j.1399-0004.2011.01748.x. Epub 2011 Aug 4. PMID 21736564
- [Background] Quarrell OW, Handley O, O'Donovan K, Dumoulin C, Ramos-Arroyo M, Biunno I, Bauer P, Kline M, Landwehrmeyer GB; European Huntington's Disease Network. Discrepancies in reporting the CAG repeat lengths for Huntington's disease. Eur J Hum Genet. 2012 Jan;20(1):20-6. doi: 10.1038/ejhg.2011.136. Epub 2011 Aug 3. PMID 21811303
- [Background] Saft C, Epplen JT, Wieczorek S, Landwehrmeyer GB, Roos RA, de Yebenes JG, Dose M, Tabrizi SJ, Craufurd D; REGISTRY Investigators of the European Huntington's Disease Network; Arning L. NMDA receptor gene variations as modifiers in Huntington disease: a replication study. PLoS Curr. 2011 Oct 4;3:RRN1247. doi: 10.1371/currents.RRN1247. PMID 21989477
- [Background] Rickards H, De Souza J, Crooks J, van Walsem MR, van Duijn E, Landwehrmeyer B, Squitieri F, Simpson SA; European Huntington's Disease Network. Discriminant analysis of Beck Depression Inventory and Hamilton Rating Scale for Depression in Huntington's disease. J Neuropsychiatry Clin Neurosci. 2011 Fall;23(4):399-402. doi: 10.1176/jnp.23.4.jnp399. PMID 22231310
- [Background] Lee JM, Ramos EM, Lee JH, Gillis T, Mysore JS, Hayden MR, Warby SC, Morrison P, Nance M, Ross CA, Margolis RL, Squitieri F, Orobello S, Di Donato S, Gomez-Tortosa E, Ayuso C, Suchowersky O, Trent RJ, McCusker E, Novelletto A, Frontali M, Jones R, Ashizawa T, Frank S, Saint-Hilaire MH, Hersch SM, Rosas HD, Lucente D, Harrison MB, Zanko A, Abramson RK, Marder K, Sequeiros J, Paulsen JS; PREDICT-HD study of the Huntington Study Group (HSG); Landwehrmeyer GB; REGISTRY study of the European Huntington's Disease Network; Myers RH; HD-MAPS Study Group; MacDonald ME, Gusella JF; COHORT study of the HSG. CAG repeat expansion in Huntington disease determines age at onset in a fully dominant fashion. Neurology. 2012 Mar 6;78(10):690-5. doi: 10.1212/WNL.0b013e318249f683. Epub 2012 Feb 8. PMID 22323755
- [Background] Henley SM, Ridgway GR, Scahill RI, Kloppel S, Tabrizi SJ, Fox NC, Kassubek J; EHDN Imaging Working Group. Pitfalls in the use of voxel-based morphometry as a biomarker: examples from huntington disease. AJNR Am J Neuroradiol. 2010 Apr;31(4):711-9. doi: 10.3174/ajnr.A1939. Epub 2009 Dec 24. PMID 20037137
- [Background] Aziz NA, Jurgens CK, Landwehrmeyer GB; EHDN Registry Study Group; van Roon-Mom WM, van Ommen GJ, Stijnen T, Roos RA. Normal and mutant HTT interact to affect clinical severity and progression in Huntington disease. Neurology. 2009 Oct 20;73(16):1280-5. doi: 10.1212/WNL.0b013e3181bd1121. Epub 2009 Sep 23. PMID 19776381
- See also: EHDN — http://www.euro-hd.net